CLINICAL TRIAL: NCT06785220
Title: The Effects of Oral Facial Facilitation and Oral Motor Therapy in Dysphagia with Spastic Cerebral Palsy
Brief Title: The Effects of Oral Facial Facilitation and Oral Motor Therapy in Dysphagia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Marwa Abd El-Mawgood Abdo Ragab, Dr, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OMT and OFF in Dysphagia
Record Dates: First submitted 2025-01-06; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Dysphagia; Spastic Cerebral Palsy (sCP)
MeSH Terms: conditions — Deglutition Disorders; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: ORAL FACIAL FACILITATION (Active Comparator): •A group will receive oral facial facilitation which included exercise for given,
  1. Brushing
  2. Vibration
  3. Manipulation (stroking and tapping)
  4. Oral motor sensory exercise (lip, tongue, swallowing exercises)
  Interventions: Other: ORAL FACIAL FACILITATION
- Group B: ORAL MOTOR THERAPY (Active Comparator): B group will receive oral motor therapy which included exercise for given,
  1. A volcano bubbles
  2. Party blower target
  3. Bubble blowing
  4. Curly straws
  Interventions: Other: ORAL MOTOR THERAPY
- Group C: ORAL FACIAL FACILITATION WITH ORAL MOROR THERAY (Active Comparator): C group will receive oral facial facilitation and oral motor therapy which included exercise for given,
  1. Brushing
  2. Vibration
  3. Manipulation (stroking and tapping)
  4. Oral motor sensory exercise (lip, tongue, swallowing exercises)
  5. A volcano bubbles
  6. Party blower target
  7. Bubble blowing
  8. Curly straws
  Interventions: Other: ORAL FACIAL FACILITATION WITH ORAL MOROR THERAY

INTERVENTIONS:
Other: ORAL FACIAL FACILITATION — A group will receive oral facial facilitation which included exercise for given,
  1. Brushing
  2. Vibration
  3. Manipulation (stroking and tapping)
  4. Oral motor sensory exercise (lip, tongue, swallowing exercises)
  Arms: Group A: ORAL FACIAL FACILITATION
Other: ORAL MOTOR THERAPY — B group will receive oral motor therapy which included exercise for given,
  1. A volcano bubbles
  2. Party blower target
  3. Bubble blowing
  4. Curly straws
  Arms: Group B: ORAL MOTOR THERAPY
Other: ORAL FACIAL FACILITATION WITH ORAL MOROR THERAY — C group will receive oral facial facilitation and oral motor therapy which included exercise for given,
  1. Brushing
  2. Vibration
  3. Manipulation (stroking and tapping)
  4. Oral motor sensory exercise (lip, tongue, swallowing exercises)
  5. A volcano bubbles
  6. Party blower target
  7. Bubble blowing
  8. Curly straws
  Arms: Group C: ORAL FACIAL FACILITATION WITH ORAL MOROR THERAY

SUMMARY:
The objective of this research is to investigate the impact of oral facial facilitation and oral motor therapy dysphagia in individuals with spastic cerebral palsy. Specifically, the study aims to:

* Evaluate changes in dysphagia and severity following a regimen of oral motor therapy and oral facial facilitation.
* Assess improvements in swallowing function, including ease of swallowing and reduction in dysphagia symptoms, after implementing oral motor therapy and oral facial facilitation.

ELIGIBILITY:
Inclusion Criteria:

* 1. Confirmed diagnosis of spastic cerebral palsy (CP) by a qualified medical professional.

  2. Participants aged 3 to 7 years, as this is a common demographic affected by spastic CP.

  3. Clinical diagnosis of dysphagia, confirmed by a speech-language pathologist or related healthcare provider.

  4. No recent significant changes in neurological status or medical condition within the last six months.

  5. Sufficient cognitive ability to follow simple instructions during therapy sessions, as assessed by a qualified professional.

  6. Parental or guardian consent obtained for participants under 18, along with assent from participants when appropriate.

  7. No recent (within the last three months) oral motor therapy interventions that could confound results.

  8. Willingness and ability of the participant to engage in therapy sessions consistently.

  9. Clearance from a physician to participate in oral motor therapy and related interventions.

Exclusion Criteria:

* 1. Diagnosis of other neurological disorders or conditions that may affect swallowing or motor skills.

  2. Serious medical conditions or comorbidities that could interfere with therapy (e.g., severe respiratory issues).

  3. Any surgical interventions affecting the oral or pharyngeal region within the last year.

  4. Concurrent participation in other clinical trials or interventions that could affect swallowing outcomes.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
functional oral intake scale | through study completion, an average of 6 months
Simplified dysphagia severity rating scale | through study completion, an average of 6 months
Eating Assessment Tool-10 | through study completion, an average of 6 months

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Furkim AM, Behlau MS, Weckx LLM. The use of cervical auscultation in tracheal aspiration in children with cerebral palsy. Rev. CEFAC. 2009;11(4):624-9.
- [Background] IOSR Journal of Dental and Medical Sciences (IOSR-JDMS) e-ISSN: 2279-0853, p-ISSN: 2279-0861.Volume 14, Issue 8 Ver. VI (Aug. 2015), PP 09-13
- [Background] Kumari P., Nikkitha E. To compare the effects of oral facial facilitation and oral motor therapy in decreasing drooling in children with spastic cerebral palsy. Int. J. Pharm. Biol. Sci. 2018;8:397-402.
- [Background] Ottenbacher K, Scoggins A, Wayland J. The effectiveness of a program of oral sensory-motor therapy with the severely and profoundly developmentally disabled. Occup Ther J Res 1981; 1: 147-60
- [Background] Walton K, Daniel AI, Mahood Q, Vaz S, Law N, Unger SL, O'Connor DL. Eating Behaviors, Caregiver Feeding Interactions, and Dietary Patterns of Children Born Preterm: A Systematic Review and Meta-Analysis. Adv Nutr. 2022 Jun 1;13(3):875-912. doi: 10.1093/advances/nmac017. PMID 35157009
- [Background] Simons A, Hamdy S. The Use of Brain Stimulation in Dysphagia Management. Dysphagia. 2017 Apr;32(2):209-215. doi: 10.1007/s00455-017-9789-z. Epub 2017 Mar 28. PMID 28353151
- [Background] Sigan SN, Uzunhan TA, Aydinli N, Eraslan E, Ekici B, Caliskan M. Effects of oral motor therapy in children with cerebral palsy. Ann Indian Acad Neurol. 2013 Jul;16(3):342-6. doi: 10.4103/0972-2327.116923. PMID 24101813
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Reilly S, Skuse D. Characteristics and management of feeding problems of young children with cerebral palsy. Dev Med Child Neurol. 1992 May;34(5):379-88. doi: 10.1111/j.1469-8749.1992.tb11449.x. PMID 1592191
- [Background] Rangarathnam B, Kamarunas E, McCullough GH. Role of cerebellum in deglutition and deglutition disorders. Cerebellum. 2014 Dec;13(6):767-76. doi: 10.1007/s12311-014-0584-1. PMID 25047686
- [Background] Pearson WG Jr, Langmore SE, Zumwalt AC. Evaluating the structural properties of suprahyoid muscles and their potential for moving the hyoid. Dysphagia. 2011 Dec;26(4):345-51. doi: 10.1007/s00455-010-9315-z. Epub 2010 Nov 11. PMID 21069388
- [Background] Parkes J, Hill N, Platt MJ, Donnelly C. Oromotor dysfunction and communication impairments in children with cerebral palsy: a register study. Dev Med Child Neurol. 2010 Dec;52(12):1113-9. doi: 10.1111/j.1469-8749.2010.03765.x. Epub 2010 Aug 31. PMID 20813020
- [Background] Park JS, Hwang NK, Kim HH, Choi JB, Chang MY, Jung YJ. Effects of lingual strength training on oropharyngeal muscles in South Korean adults. J Oral Rehabil. 2019 Nov;46(11):1036-1041. doi: 10.1111/joor.12835. Epub 2019 Jul 2. PMID 31206763
- [Background] Pakula AT, Van Naarden Braun K, Yeargin-Allsopp M. Cerebral palsy: classification and epidemiology. Phys Med Rehabil Clin N Am. 2009 Aug;20(3):425-52. doi: 10.1016/j.pmr.2009.06.001. PMID 19643346
- [Background] Min KC, Seo SM, Woo HS. Oral-motor facilitation technique (OMFT): Part I-Theoretical Base and Basic Concept. Therapeutic Sci Rehabilitation. 2021;10(1):37-52. https://doi.org/10.22683/tsnr.2021.10.1.037
- [Background] Min KC, Seo SM, Woo HS. Oral-motor facilitation technique (OMFT): Part II-Conceptual Hierarchy and Key Point Technique. Therapeutic Sci Rehabilitation. 2021;10(1):53-61. https://doi.org/10.22683/tsnr.2021.10.1.053.
- [Background] Makris T, Dorstyn D, Crettenden A. Quality of life in children and adolescents with cerebral palsy: a systematic review with meta-analysis. Disabil Rehabil. 2021 Feb;43(3):299-308. doi: 10.1080/09638288.2019.1623852. Epub 2019 Jun 10. PMID 31180733
- [Background] Li XL, Liu Y, Liu M, Yang CY, Yang QZ. Early Premature Infant Oral Motor Intervention Improved Oral Feeding and Prognosis by Promoting Neurodevelopment. Am J Perinatol. 2020 May;37(6):626-632. doi: 10.1055/s-0039-1685448. Epub 2019 Apr 23. PMID 31013539
- [Background] Engle RP, Canner GC. Proprioceptive Neuromuscular Facilitation (PNF) and Modified Procedures for Anterior Cruciate Ligament (ACL) Instability. J Orthop Sports Phys Ther. 1989;11(6):230-6. doi: 10.2519/jospt.1989.11.6.230. PMID 18796905
- [Background] Graham HK, Rosenbaum P, Paneth N, Dan B, Lin JP, Damiano DL, Becher JG, Gaebler-Spira D, Colver A, Reddihough DS, Crompton KE, Lieber RL. Cerebral palsy. Nat Rev Dis Primers. 2016 Jan 7;2:15082. doi: 10.1038/nrdp.2015.82. PMID 27188686
- [Background] Gisel EG. Oral-motor skills following sensorimotor intervention in the moderately eating-impaired child with cerebral palsy. Dysphagia. 1994 Summer;9(3):180-92. doi: 10.1007/BF00341263. PMID 8082327
- [Background] Chaleat-Valayer E, Porte M, Buchet-Poyau K, Roumenoff-Turcant F, D'Anjou MC, Boulay C, Bernard JC, Touzet S. Management of drooling in children with cerebral palsy: A French survey. Eur J Paediatr Neurol. 2016 Jul;20(4):524-31. doi: 10.1016/j.ejpn.2016.04.010. Epub 2016 Apr 22. PMID 27155820
- [Background] Owen SE, Stern ML. Management of drooling in cerebral palsy: three single case studies. Int J Rehabil Res. 1992;15(2):166-9. doi: 10.1097/00004356-199206000-00011. No abstract available. PMID 1526706
- [Background] Frakking TT, Chang AB, O'Grady KF, David M, Walker-Smith K, Weir KA. The Use of Cervical Auscultation to Predict Oropharyngeal Aspiration in Children: A Randomized Controlled Trial. Dysphagia. 2016 Dec;31(6):738-748. doi: 10.1007/s00455-016-9727-5. Epub 2016 Jul 11. PMID 27402004
- [Background] Dawes C, Pedersen AM, Villa A, Ekstrom J, Proctor GB, Vissink A, Aframian D, McGowan R, Aliko A, Narayana N, Sia YW, Joshi RK, Jensen SB, Kerr AR, Wolff A. The functions of human saliva: A review sponsored by the World Workshop on Oral Medicine VI. Arch Oral Biol. 2015 Jun;60(6):863-74. doi: 10.1016/j.archoralbio.2015.03.004. Epub 2015 Mar 10. PMID 25841068
- [Background] Clancy KJ, Hustad KC. Longitudinal changes in feeding among children with cerebral palsy between the ages of 4 and 7 years. Dev Neurorehabil. 2011;14(4):191-8. doi: 10.3109/17518423.2011.568467. PMID 21732803
- [Background] Calis EA, Veugelers R, Sheppard JJ, Tibboel D, Evenhuis HM, Penning C. Dysphagia in children with severe generalized cerebral palsy and intellectual disability. Dev Med Child Neurol. 2008 Aug;50(8):625-30. doi: 10.1111/j.1469-8749.2008.03047.x. PMID 18754902
- [Background] Burkhead LM, Sapienza CM, Rosenbek JC. Strength-training exercise in dysphagia rehabilitation: principles, procedures, and directions for future research. Dysphagia. 2007 Jul;22(3):251-65. doi: 10.1007/s00455-006-9074-z. Epub 2007 Apr 25. PMID 17457549
- [Background] Boel L, Pernet K, Toussaint M, Ides K, Leemans G, Haan J, Van Hoorenbeeck K, Verhulst S. Respiratory morbidity in children with cerebral palsy: an overview. Dev Med Child Neurol. 2019 Jun;61(6):646-653. doi: 10.1111/dmcn.14060. Epub 2018 Oct 15. PMID 30320434
- [Background] Blair E, Watson L, Badawi N, Stanley FJ. Life expectancy among people with cerebral palsy in Western Australia. Dev Med Child Neurol. 2001 Aug;43(8):508-15. doi: 10.1017/s0012162201000949. PMID 11508916
- [Background] Bax M, Tydeman C, Flodmark O. Clinical and MRI correlates of cerebral palsy: the European Cerebral Palsy Study. JAMA. 2006 Oct 4;296(13):1602-8. doi: 10.1001/jama.296.13.1602. PMID 17018805
- [Background] Kaviyani Baghbadorani M, Soleymani Z, Dadgar H, Salehi M. The effect of oral sensorimotor stimulations on feeding performance in children with spastic cerebral palsy. Acta Med Iran. 2014;52(12):899-904. PMID 25530052
- [Background] Arvedson J, Clark H, Lazarus C, Schooling T, Frymark T. The effects of oral-motor exercises on swallowing in children: an evidence-based systematic review. Dev Med Child Neurol. 2010 Nov;52(11):1000-13. doi: 10.1111/j.1469-8749.2010.03707.x. PMID 20497451